CLINICAL TRIAL: NCT07263100
Title: Comparative Study Between Intralesional Corticosteroid Injection Alone and Combined Intralesional Corticosteroid Injection With Either Long-pluse Nd YAG or Erbium Yag for Treating Hypertrophic or Keloid Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somdech Phra Nangchao Sirikit Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: RP009/66
Record Dates: First submitted 2024-11-12; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Hypertrophic Scar; Keloid; Laser
Keywords: Hypertrophic scar; Keloid; Laser
MeSH Terms: conditions — Cicatrix, Hypertrophic; Keloid | interventions — Triamcinolone Acetonide; Lasers, Solid-State

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Keloidal scar (Active Comparator): Randomly assigned keloid scar to each intervention (IL KA)
  Interventions: Drug: Triamcinolone acetonide injection
- Keloidal scar 2 (Experimental): Randomly assigned keloid scar to each intervention (IL KA + ND YAG)
  Interventions: Device: Fotona dynamis: Long pulse Nd YAG + Er YAG laser
- Keloidal scar 3 (Experimental): Randomly assigned keloid scar to each intervention (ILKA + Er YAG)
  Interventions: Device: Fotona Dynamis: Long pulse Nd YAG + Er YAG laser

INTERVENTIONS:
Drug: Triamcinolone acetonide injection — Long-pulse ND YAG and Erbium YAG laser device: Fotona Dynamis
  Arms: Keloidal scar
Device: Fotona dynamis: Long pulse Nd YAG + Er YAG laser — Intralesional corticosteroid injection combine with long-pulse Neodynium-doped Yttrium Aluminium Garnet Laser (Nd-YAG) (IL KA + ND YAG)
  Arms: Keloidal scar 2
Device: Fotona Dynamis: Long pulse Nd YAG + Er YAG laser — Intralesional corticosteroid injection combine with Erbium Yttrium Aluminium Garnet Laser (Er-YAG) (IL KA + Er YAG)
  Arms: Keloidal scar 3

SUMMARY:
To compare the effectiveness of hypertrophic or keloid scar treatment with either intralesional corticosteroid injection alone or combined intralesional corticosteroid injection with either long-pulse ND YAG or Erbium YAG

ELIGIBILITY:
Inclusion Criteria:

* Individual with hypertrophic or keloid scars on any location
* Size of hypertrophic or keloid scars not larger than 20 cms in diameter

Exclusion Criteria:

* Any topical or procedural treatment on scar in last 6 months
* Current corticosteroid use
* Bleeding disorders or coagulopathies
* Pregnancy or nursing
* Chronic kidney diseases
* Chronic liver diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Vancouver scar scale | 5 months
  Vancouver scar scale to evaluate scar severity of keloid scar assessing 4 variations including vascularity, pigmentation, pliability, height scoring range from 0-13 (the more scores resembling the more severity)

SECONDARY OUTCOMES:
Japan Scar Workshop Scar Scale | 5 months
  Japan Scar Workshop Scar Scale to evaluate scar severity of keloid scar assessing 2 main domains (risk factors and presenting symptoms) by 2 tables
  1. Classification scoring range 0-5 = matured scars 6-15 = hypertrophic scars 16-25 = keloids
  2. Evaluation for treatment & follow ups scoring range from 0-18 (the more scores resembling the more severity)

CONTACTS AND LOCATIONS:
Locations (1):
- Somdech Phra Nangchao Sirikit Hospital, Sattahip, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient demographic data and scar characteristics, severity can be shared upon requests
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1st July 2025 - 31st Dec 2025
Access Criteria: Patient demographic data and scar characteristics, severity can be shared upon requests by emailing to the main researchers and asking for permission
URL: https://drive.google.com/drive/folders/13Ki4kcn2QTHplGT0HjuEiCUlJJplC7dv?usp=drive_link

REFERENCES:
- [Background] Park JH, Jeong JW, Park JU. Efficacy of Nd:YAG Laser and Intralesional Triamcinolone Injection Combination Therapy in the Postoperative Management of Keloids. Aesthetic Plast Surg. 2025 Jan;49(2):576-583. doi: 10.1007/s00266-024-04433-z. Epub 2024 Oct 7. PMID 39373734